CLINICAL TRIAL: NCT02869347
Title: Recombinant Human C1 Esterase Inhibitor (Conestat Alfa) in the Prevention of Contrast-induced Nephropathy in High-risk Subjects (PROTECT): a Randomized, Placebo-controlled, Double-blind Single-center Trial
Brief Title: Recombinant Human C1 Esterase Inhibitor in the Prevention of Contrast-induced Nephropathy in High-risk Subjects
Acronym: PROTECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Pharming Technologies B.V. (Industry); Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BASEC 2016-01112
Record Dates: First submitted 2016-08-12; First posted 2016-08-16 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Acute Kidney Injury
Keywords: recombinant C1 esterase inhibitor; acute kidney injury; coronary angiography; contrast media; Conestat alfa; inflammation
MeSH Terms: conditions — Acute Kidney Injury; Inflammation | interventions — conestat alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conestat alfa (Active Comparator): Intravenous injection of Conestat alfa, for patients less than 84kg at a dose of 50 U/kg, and for patients of 84kg body weight or greater at a dose of 4200 U (2 vials, each diluted in 14ml sterile water).
  Interventions: Drug: Conestat alfa
- Sodium chloride 0.9% (Placebo Comparator): Intravenous injection of sodium chloride 0.9%.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Conestat alfa — Two intravenous injections (over 5 minutes) of Conestat alfa immediately pre-procedure (elective coronary angiography) and 4 hours later; for patients less than 84kg at a dose of 50 U/kg, and for patients of 84kg body weight or greater at a dose of 4200 U.
  Other Names: recombinant human C1 esterase inhibitor
  Arms: Conestat alfa
Drug: Sodium chloride 0.9% — Two intravenous injections of sodium chloride 0.9% (maximum 28 ml, matching the respective amount of the Conestat alfa arm) immediately pre-procedure (elective coronary angiography) and 4 hours later.
  Other Names: isotonic (normal) saline
  Arms: Sodium chloride 0.9%

SUMMARY:
Iodinated contrast media have been causally linked to acute kidney injury known as contrast-induced nephropathy (CIN), which is the consequence of CM-induced local renal ischemia and direct toxic effects. Conestat alfa (recombinant human C1 esterase inhibitor) has been shown to decrease renal ischemic damage in experimental models of renal ischemia.

The Recombinant Human C1 Esterase Inhibitor in the Prevention of Contrast-induced Nephropathy in High-risk Subjects (PROTECT) Study is a randomized, placebo-controlled, double-blind single-center trial that will assess the effect of prophylactic administration of Conestat alfa on the degree of acute kidney injury subjects undergoing elective coronary angiography. Patient with an estimated glomerular filtration rate <=50 ml/min/1.73 m2 and at least one additional risk factor for CIN will be enrolled and randomly assigned to 1) Conestat alfa at 50 U/kg given as intravenous injection immediately before and 4 hours after coronary angiography or 2) placebo (sodium chloride). All patients will receive standard intravenous hydration with isotonic saline. Surrogate markers of kidney injury will be assessed over a 48 hours time period. Patients will be followed for cardiovascular and renal events over 12 weeks.

The primary outcome measure is peak change in urinary Neutrophil gelatinase-associated lipocalin within 48 hours after elective coronary angiography.

DETAILED DESCRIPTION:
Iodinated contrast media (CM) are an essential component of contemporary imaging and interventional studies. Although CM are generally well tolerated, they have been causally linked to acute kidney injury known as contrast-induced nephropathy (CIN), the third leading cause of acute kidney injury in hospitalized patients. Preexisting renal impairment, diabetes mellitus, advanced age, congestive heart failure, or large volumes and repeated use of CM have been identified as risk factors for CIN. CIN is the consequence of CM-induced local renal ischemia in combination with direct toxic effects to renal tubular cells. Subsequent inflammation may cause further tissue damage in the reperfusion period. Apart from intravenous hydration preventive strategies for CIN are lacking.

The complement system consists of several circulating proteins that are implicated in the first-line defence against pathogens and in the removal of dying cells. Following renal ischemia activation of the lectin pathway of complement in particular has been associated with local tissue damage in the kidney. Conestat alfa is a recombinant human C1 esterase inhibitor, which inhibits activation of the complement system and is licensed in Europe and USA for the treatment of a hereditary condition (hereditary angioedema). Conestat alfa markedly reduced tissue damage in experimental models of renal ischemia and reperfusion injury, but has not been investigated in human ischemia.

The Recombinant Human C1 Esterase Inhibitor in the Prevention of Contrast-induced Nephropathy in High-risk Subjects (PROTECT) Study is a randomized, placebo-controlled, double-blind single-center trial that will assess the effect of prophylactic administration of Conestat alfa on the degree of acute kidney injury subjects undergoing elective coronary angiography. Patient with an estimated glomerular filtration rate <=50 ml/min/1.73 m2 and at least one additional risk factor for CIN will be enrolled and randomly assigned to 1) Conestat alfa at 50 U/kg given as intravenous injection immediately before and 4 hours after coronary angiography or 2) placebo (sodium chloride). All patients will receive standard intravenous hydration with isotonic saline. Surrogate markers of kidney injury including serum creatinine and cystatin C and urinary Neutrophil gelatinase-associated lipocalin and TIMP2 * Insulin-like growth factor-binding protein 7 (IGFBP7) will be assessed over a 48 hours time period. In addition, increases in troponin T, a marker of cardiac damage, will be assessed. Patients will be followed for thromboembolic, anaphylactic and a composite endpoint of cardiovascular and renal events over a 12 week period.

The primary outcome measure is peak change in urinary Neutrophil gelatinase-associated lipocalin within 48 hours after elective coronary angiography.

Total hydration and contrast media volume will be recorded. Serum C1 esterase inhibitor levels immediately before and 10 minutes after administration of Conestat alfa or placebo will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) of <50 ml/min/1.73m2
* At least one of the following risk factors: diabetes mellitus, age at least 75 years, anemia (baseline hematocrit value less or equal 39% for men and less or equal 36% for women), congestive heart failure class III or IV by New York Heart Association classification, history of pulmonary edema.

Exclusion Criteria:

* Contraindications to the class of drugs under study (C1 esterase inhibitors), e.g. known hypersensitivity or allergy to class of drugs or the investigational product
* History of allergy to rabbits
* Current treatment with N-acetylcysteine, sodium bicarbonate, fenoldopam, mannitol (not applicable to mannitol serving as excipient in other medical drugs), dopamine or theophylline
* Women who are pregnant or breast feeding
* Multiple myeloma
* Acute decompensated heart failure (requiring hospital admission and treatment with supplemental oxygen, diuretics and/or vasodilator therapy) within two weeks prior to the date of coronary angiography
* Acute myocardial infarction (ST elevation or non-ST elevation myocardial infarction) within two weeks prior to the date of coronary angiography
* Dialysis
* Exposure to iodinated contrast media within seven days prior to the date of coronary angiography.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigators and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Peak change from baseline of urinary Neutrophil gelatinase-associated lipocalin | within 48 hours after contrast exposure
  measured at baseline, 4, 24 and 48 hours

SECONDARY OUTCOMES:
Development of contrast-induced nephropathy | within 48 hours after contrast exposure
  contrast-induced nephropathy is defined as serum creatinine increase of at least 25% or 44micromol/L within 48 hours after coronary angiography
Cystatin C increase of at least 10% | within 24 hours after contrast exposure
  measured at baseline and 24 hours
increase in troponin T | within 24 hours after contrast exposure
  measured at baseline, 4 and 24 hours
Peak change from baseline of urinary TIMP2 * IGFBP7 | within 48 hours after contrast exposure
  measured at baseline, 4, 24 and 48 hours

OTHER OUTCOMES:
Composite cardiovascular and renal outcome | within 12-weeks after first intervention
  defined as death, unstable angina/acute coronary syndrome, hospitalization for heart or renal failure, or hemodialysis
Thromboembolic events | within 12-weeks after first intervention
  defined as symptomatic deep vein thrombosis or pulmonary embolism
Anaphylactic reaction | within 24 hours after first intervention
  defined as acute onset of an illness involving the skin and/or mucosa and either respiratory compromise or reduced blood pressure/evidence of end-organ malperfusion
C1 inhibitor serum concentration | Baseline and 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michael Osthoff, M.D., Principal Investigator — University Hospital Basel, Department of Infectious Diseases
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Panagiotou A, Trendelenburg M, Heijnen IAFM, Moser S, Bonati LH, Breidthardt T, Fahrni G, Kaiser C, Jeger R, Osthoff M. A Randomized Trial of Recombinant Human C1-Esterase-Inhibitor in the Prevention of Contrast-Induced Kidney Injury. JACC Cardiovasc Interv. 2020 Apr 13;13(7):833-842. doi: 10.1016/j.jcin.2019.11.021. Epub 2020 Mar 11. PMID 32171721